CLINICAL TRIAL: NCT05665946
Title: Acute Intestinal Ischaemia: the Preoperative Diagnostic Approach
Brief Title: Acute Intestinal Necrosis- the Preoperative Diagnostic Approach
Acronym: AIN
Status: Completed | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, David Straarup, Principal Investigator, Aalborg University Hospital
Other Study IDs: AalborgAIN
Record Dates: First submitted 2022-12-09; First posted 2022-12-27 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Acute Mesenteric Ischemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Full blood samples drawn just after inclusion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AIN patients: Surgical verified AIN patients. A blood sample is drawn just after inclusion and stored for later analysis.
  Interventions: Diagnostic Test: Blood sample analysis
- Controls.: Non-AIN patients. A blood sample is drawn just after inclusion and stored for later analysis.
  Interventions: Diagnostic Test: Blood sample analysis

INTERVENTIONS:
Diagnostic Test: Blood sample analysis — Analysis of proposed biomarkers.

SUMMARY:
To investigate a number of blood based parameters in patients with intestinal ischaemia compared to patients with other acute abdominal diseases.

DETAILED DESCRIPTION:
Intestinal ischemia is a life-threatening condition defined by interrupted blood supply to the intestinal tissue. Primary and secondary ischemia is obstruction of blood-supply due to vascular and extra-vascular pathology, respectively.

Early diagnosis and treatment are critical to save the ischemic bowel. Clinical findings of secondary intestinal ischaemia are related to the underlying cause e.g. vomiting and palpable hernia. Abdominal computed tomography (CT) can effectively visualize the causes. In contrast, the diagnosis of primary intestinal ischemia is often delayed due to the absence of specific clinical findings. Primary intestinal ischemia is visualized with CT ateriography, revealing mesentery arterial obstruction. However, in the acute setting a non-arterial phase CT is often performed but the findings are unspecific in the early stages and the pattern of findings which could indicate primary ischemia are not well understood. In primary and secondary ischemia, standard blood-based parameters are inconsistently elevated and highly unspecific. Newer blood-based parameters such as D-lactate has been proposed as ischaemic markers. D-lactate is produced by bacteria in the bowel lumen and translocation through a damaged bowel wall makes it a potential marker of intestinal ischemia.

A case-control-study of all acute admitted patients with abdominal pain in Aalborg, Denmark in the mentioned time range. The sensitivity and specificity of potiential biomarkers in a blood sample at time of admission as a marker of intestinal ischaemia will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Referred to The Department of Gastrointestinal Surgery, Aalborg University Hospital.

Exclusion Criteria:

* Children

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Referred patient from the whole uptake area whic is 590.000 inhabitans for regional hospital functions.
Sampling Method: Non-Probability Sample
Enrollment: 2958 (Actual)
Dates: Start 2015-01-06 (Actual); Primary Completion 2019-03-24 (Actual); Study Completion 2019-03-24 (Actual)

PRIMARY OUTCOMES:
D-lactate | 2015-2019, Just after inclusion
  Measurement of baseline level of D-lactate as a predictor of AIN
I-FABP | 2015-2019, Just after inclusion
  Measurement of baseline level of I-FABP as a predictor of AIN.
Endothelin-1 | 2015-2019, Just after inclusion
  Measurement of baseline level of Endothelin-1 as a predictor of AIN
L-lactate | 2015-2019, Just after inclusion
  Measurement of baseline level of L-lactate as a predictor of AIN

CONTACTS AND LOCATIONS:
Overall Officials: David Straarup, MD, Principal Investigator — Dept. of Gastrointestinal Surgery, Aalborg University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adaba F, Askari A, Dastur J, Patel A, Gabe SM, Vaizey CJ, Faiz O, Nightingale JM, Warusavitarne J. Mortality after acute primary mesenteric infarction: a systematic review and meta-analysis of observational studies. Colorectal Dis. 2015 Jul;17(7):566-77. doi: 10.1111/codi.12938. PMID 25739990
- [Background] Assadian A, Assadian O, Senekowitsch C, Rotter R, Bahrami S, Furst W, Jaksch W, Hagmuller GW, Hubl W. Plasma D-lactate as a potential early marker for colon ischaemia after open aortic reconstruction. Eur J Vasc Endovasc Surg. 2006 May;31(5):470-4. doi: 10.1016/j.ejvs.2005.10.031. Epub 2005 Dec 22. PMID 16376117
- [Background] Block T, Nilsson TK, Bjorck M, Acosta S. Diagnostic accuracy of plasma biomarkers for intestinal ischaemia. Scand J Clin Lab Invest. 2008;68(3):242-8. doi: 10.1080/00365510701646264. PMID 17934974
- [Background] Corcos O, Nuzzo A. Gastro-intestinal vascular emergencies. Best Pract Res Clin Gastroenterol. 2013 Oct;27(5):709-25. doi: 10.1016/j.bpg.2013.08.006. Epub 2013 Sep 5. PMID 24160929
- [Background] Dohle DS, Bestendonk C, Petrat F, Tsagakis K, Wang M, Strucksberg KH, Canbay A, Jakob H, de Groot H. Serum markers for early detection of patients with mesenteric ischemia after cardiac surgery. Innov Surg Sci. 2018 Nov 30;3(4):277-283. doi: 10.1515/iss-2018-0035. eCollection 2018 Dec. PMID 31579792
- [Background] Nuzzo A, Guedj K, Curac S, Hercend C, Bendavid C, Gault N, Tran-Dinh A, Ronot M, Nicoletti A, Bouhnik Y, Castier Y, Corcos O, Peoc'h K; SURVI (Structure d'URgences Vasculaires Intestinales) Research Group (French Intestinal Stroke Center). Accuracy of citrulline, I-FABP and D-lactate in the diagnosis of acute mesenteric ischemia. Sci Rep. 2021 Sep 23;11(1):18929. doi: 10.1038/s41598-021-98012-w. PMID 34556697
- [Background] Tilsed JV, Casamassima A, Kurihara H, Mariani D, Martinez I, Pereira J, Ponchietti L, Shamiyeh A, Al-Ayoubi F, Barco LA, Ceolin M, D'Almeida AJ, Hilario S, Olavarria AL, Ozmen MM, Pinheiro LF, Poeze M, Triantos G, Fuentes FT, Sierra SU, Soreide K, Yanar H. ESTES guidelines: acute mesenteric ischaemia. Eur J Trauma Emerg Surg. 2016 Apr;42(2):253-70. doi: 10.1007/s00068-016-0634-0. PMID 26820988
- [Background] Reintam Blaser A, Forbes A, Bjorck M. Acute mesenteric ischaemia. Curr Opin Crit Care. 2022 Dec 1;28(6):702-708. doi: 10.1097/MCC.0000000000000972. Epub 2022 Aug 10. PMID 35950719
- [Derived] Straarup D, Gotschalck KA, Christensen PA, Krarup H, Lundbye-Christensen S, Handberg A, Thorlacius-Ussing O. Exploring I-FABP, endothelin-1 and L-lactate as biomarkers of acute intestinal necrosis: a case-control study. Scand J Gastroenterol. 2023 Jul-Dec;58(12):1359-1365. doi: 10.1080/00365521.2023.2229930. Epub 2023 Jul 4. PMID 37403410